CLINICAL TRIAL: NCT00324649
Title: Pilot Phase IV, Multicenter, Randomized, Open-label and Controlled Study to Assess the Evolution of Peripheral Body Fat Distribution After Switching From Zidovudine Containing Backbone to Truvada in HIV-1-infected Patients on HAART (RECOMB Study).
Brief Title: Peripheral Body Fat Distribution After Switching Zidovudine and Lamivudine to Truvada
Acronym: RECOMB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-ES-164-0154
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2009-05-20 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: HIV-1
Keywords: HIV-1
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Truvada (Experimental): Truvada + NNRTI or PI.
  Interventions: Drug: Truvada
- Zidovudine/lamivudine (Active Comparator): Zidovudine/lamivudine + NNRTI or PI.
  Interventions: Drug: Zidovudine/lamivudine

INTERVENTIONS:
Drug: Truvada — Truvada once daily with continuation of the current NNRTI or PI at randomization.
  Arms: Truvada
Drug: Zidovudine/lamivudine — Continuation of the zidovudine + lamivudine containing regimen plus the current NNRTI or PI at randomization.
  Arms: Zidovudine/lamivudine

SUMMARY:
This study evaluated changes in body fat distribution in human immunodeficiency virus type 1 (HIV-1) infected participants who either switched from a zidovudine- plus lamivudine- containing highly active antiretroviral therapy (HAART) regimen to a regimen containing Truvada® (a fixed-dose combination tablet of emtricitabine [FTC, 200 mg] and tenofovir disoproxil fumarate [TDF, 300 mg]) or who remained on a zidovudine- plus lamivudine-containing regimen. Subjects continued their protease inhibitor (PI) or nonnucleoside reverse transcriptase inhibitor (NNRTI).

DETAILED DESCRIPTION:
Standard care for the treatment of HIV infection involves the use of a combination of three antiretroviral drugs. The initial recommended regimen in antiretroviral-naive patients according to therapeutic guidelines of the US Department of Health and Human Resources (DHHS) includes two nucleoside reverse transcriptase inhibitors (NRTIs) and a third drug from another class (PI or NRTI).

The use of nucleoside analogues, especially stavudine and zidovudine, is associated with untoward side effects, including lipodystrophy hepatic steatosis/lactic acidosis syndrome, peripheral neuropathy, and anemia. However, Truvada has a low potential for both mitochondrial toxicity and fat distribution disturbances.

As described in the Consensus Document of the Spanish Group for the Study of AIDS (GESIDA), and the AIDS National Plan from the Spanish Ministry of Health "Recommendations on metabolic alterations and body fat distribution", studies should focus on the evaluation of body fat disturbances after antiretroviral drug substitutions, based on the basic assumption of virologic control of the patient and equivalence in potency of the new drug regarding virological control. In addition, studies based on selective substitution of antiretroviral drugs in HIV-1 infected patients under virological control, are recommended in the European Medicines Agency (EMA) in the "Guideline on the clinical development of medicinal products for the treatment of HIV infection".

In this study, stable, virologically controlled, HIV-1 infected participants receiving antiretroviral regimens containing zidovudine and lamivudine were randomized to switch to Truvada or to stay on their zidovudine- plus lamivudine-containing regimen. Participants in both groups continued the third drug of their antiretroviral regimen (either an NNRTI or PI). Changes in limb fat in the two groups were assessed using dual-energy x-ray absorptiometry (DEXA).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by confirmed positive HIV-1 antibody test and/or positive polymerase chain reaction for HIV-1 ribonucleic acid (RNA).
* Adult patients (over 18 years of age).
* Current HAART regimen containing zidovudine + lamivudine at usual doses for at least 6 months.
* Viral load < 50 copies/mL on the last two consecutive determinations, under zidovudine + lamivudine containing HAART regimen.
* For women of childbearing potential, negative urine pregnancy test at screening visit.
* Agreement to take part in the study and sign the informed consent.
* Patients on lipid lowering treatment were allowed to participate in the study only if the lipid-lowering treatment (either statins or fibrates) was stable for at least 8 weeks prior to screening and it was not expected to change during the first 3 months of the study.

Exclusion Criteria:

* Patients on current FTC or TDF therapy.
* Patients with previous history of virological failure on an FTC or TDF-containing regimen.
* Patients receiving a non-registered antiretroviral drug.
* Patients receiving a triple-nucleoside antiretroviral combination.
* Hypersensitivity to one of the components of the dosage forms of TDF or FTC, or previous history of intolerance to one of those drugs.
* Known history of drug abuse or chronic alcohol consumption
* Women who were pregnant or breast feeding, or female of childbearing potential who did not use an adequate method of contraception according to the investigator's judgment.
* Active opportunistic infection or documented infection within the previous 4 weeks.
* Documented active malignant disease (excluding Kaposi sarcoma limited to the skin).
* Renal disease with creatinine clearance < 50 mL/min.
* Concomitant use of nephrotoxic or immuno-suppressive drugs which could not be stopped without affecting the safety of the patient.
* Receiving on-going therapy with systemic corticosteroids, Interleukin-2 or chemotherapy.
* Patients who were not to be included in the study according to the investigator's criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ferrer, Study Director — Gilead Sciences, S.L.
Locations (1):
- Gilead Sciences, S.L., Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Truvada: Truvada + nonnucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI).
- Zidovudine/Lamivudine: Zidovudine/lamivudine + nonnucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI).
Period: Overall Study
Arm/Group | Truvada | Zidovudine/Lamivudine
Started | 39 | 41
Completed | 37 | 36
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Truvada | Zidovudine/Lamivudine | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10.6) | 44 (7.4) | 44 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15.0
  Male | 28 | 37 | 65.0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 36 | 38 | 74.0
  Black, of African heritage | 1 | 2 | 3.0
  Asian | 1 | 0 | 1.0
  Other | 1 | 1 | 2.0
Region of Enrollment [Number; unit: participants]
  Spain | 39 | 41 | 80.0
HIV-1 RNA Level [Number; unit: Participants]
  < 50 copies/mL | 38 | 39 | 77.0
  50 to < 400 copies/mL | 1 | 2 | 3.0
Cluster determinant 4 (CD4) cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 655.0 [505.0 to 789.0] | 504.0 [363.0 to 756.0] | 600.5 [420.0 to 760.5]
Total limb fat [Median (Full Range); unit: grams (g)] — Measured using dual-energy x-ray absorptiometry (DEXA). Total limb fat is the sum of the left arm, right arm, left leg, and right leg.
  grams (g) | 3565 [511 to 15932] | 3589 [903 to 28155] | 3589 [511 to 28155]
Years on zidovudine (AZT)/lamivudine (3TC) [Median (Inter-Quartile Range); unit: Years] | 5.8 [4.2 to 7.2] | 6.2 [4.7 to 7.2] | 5.9 [4.6 to 7.2]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Limb Fat at Week 48
Description: Limb fat was measured by DEXA. Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Number of participants analyzed is those with baseline and post-baseline DEXA data. Last post-baseline observation carried forward (LOCF) method was used if the Week 48 limb fat value was missing.
Measure: Median (Inter-Quartile Range); unit: grams (g)
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 38 | 38
grams (g) | 392 [-102 to 1056] | -257 [-751 to 148]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; Null Hypothesis: changes from baseline in the two treatment groups are equal. Alternative Hypothesis: changes from baseline in the two treatment groups are different (two sided); Test type: Superiority or Other; p = 0.0014, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

2. Secondary Outcome: Change From Baseline in the Mitochondrial DNA/Nuclear DNA Ratio (Oral Mucosa)
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 34 | 35
Ratio | 62.0 [20.0 to 212.0] | 97.0 [20.0 to 197.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9713, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

3. Secondary Outcome: Change From Baseline in the Mitochondrial DNA/Nuclear DNA Ratio (Lymphocytes)
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 36 | 35
Ratio | 36.0 [2.0 to 89.5] | 43.0 [1.0 to 72.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9725, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

4. Secondary Outcome: Change From Baseline in Lactate Concentration
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 27 | 30
mmol/L | -0.23 [-0.55 to 0.00] | 0.09 [-0.12 to 0.43]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0078, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

5. Secondary Outcome: Percentage of Days for Which Participants Were Compliant With Study Drug
Description: Compliance = [1 - [(sum of days with a missed dose [per Question 6 study medication assessment questionnaire (SMAQ)])/(sum of days between SMAQ visits)]] *100 for visits with SMAQ data. An assessable visit is one where the number of missed days was reported [Question 6] and the number of days between SMAQ visits could be calculated.
Time Frame: Baseline to Week 72
Population: Treated participants.
Measure: Median (Inter-Quartile Range); unit: Percentage of days with compliance
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 39 | 41
Percentage of days with compliance | 100.0 [99.8 to 100.0] | 100.0 [99.6 to 100.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; Null Hypothesis: percentages of days with compliance in the two treatment groups are equal. Alternative Hypothesis: percentages of days with compliance in the two treatment groups are different (two sided); Test type: Superiority or Other; p = 0.6984, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

6. Secondary Outcome: Percentage of Participants Who Maintain Confirmed HIV-1 RNA < 50 Copies/mL
Time Frame: 48 weeks
Population: Treated participants. Missing values were treated as failure (i.e., as HIV-1 RNA greater than or equal to 50 copies/mL).
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 39 | 41
Percentage of participants | 92.3 | 78.0
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; Null Hypothesis: treatment is not associated with the observed virologic response. Alternative Hypothesis: treatment is associated with the observed virologic response; Test type: Superiority or Other; p = 0.1165, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made; Mean Difference (Net) = 14.3, 95% CI [-0.9 to 29.4] — The difference is for Truvada minus zidovudine/lamivudine. The 95% confidence interval on the mean difference between treatment groups is based on the normal approximation

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA > 50 and < 400 Copies/mL
Time Frame: 48 weeks
Population: Treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 39 | 41
Percentage of participants | 0 | 5

8. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as two consecutive HIV RNA values > 400 copies/mL.
Time Frame: 48 weeks
Population: Treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 39 | 41
Percentage of participants | 0 | 0

9. Secondary Outcome: Change From Baseline in Cluster Determinant 4 (CD4) Cell Count
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 36 | 34
cells/mm^3 | 60.5 [-6.5 to 159.0] | 9.0 [-61.0 to 106.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0789, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

10. Secondary Outcome: Change From Baseline in Fasting Serum Triglycerides
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 34 | 31
mg/dL | 1.5 [-31.0 to 17.0] | 4.0 [-44.0 to 40.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9633, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

11. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 34 | 31
mg/dL | 4.5 [-12.0 to 12.0] | 1.0 [-19.0 to 21.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9686, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

12. Secondary Outcome: Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL)
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 29 | 27
mg/dL | 7.0 [-9.4 to 15.6] | 5.0 [-14.0 to 16.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6638, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were performed; No adjustments were made

13. Secondary Outcome: Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL)
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 31 | 28
mg/dL | -2.0 [-7.0 to 2.0] | 2.0 [-7.0 to 7.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2907, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

14. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 36 | 33
g/dL | 0.9 [0.0 to 1.2] | 0.3 [-0.5 to 0.7]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0072, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

15. Secondary Outcome: Percent Change From Baseline in Hematocrit
Description: Change = Week 48 value minus baseline value expressed as median percent change.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: Percent change in hematocrit
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 36 | 33
Percent change in hematocrit | 2.7 [1.5 to 4.3] | 1.0 [-0.9 to 2.0]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

16. Secondary Outcome: Change From Baseline in Waist Circumference/Hip Circumference Ratio
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: Treated participants. Missing values were excluded. Assessment of waist and hip circumference was added to the study schedule via protocol amendment part way through the study. This resulted in small numbers of subjects having data available for this analysis.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 28 | 25
Ratio | -0.01 [-0.03 to 0.02] | 0.01 [-0.01 to 0.04]
Statistical Analysis 1: Comparison: Truvada vs Zidovudine/Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1785, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

17. Secondary Outcome: Percentage of Participants With Any Adverse Event
Description: Participants with treatment-emergent adverse events were analyzed. Adverse events were defined as any untoward medical occurrence in a clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with study treatment, and were categorized using the Medical Dictionary for Regulatory Activities (MedDRA) Version 11.
  Treatment-emergent adverse events were events that met one of the following criteria:
  * Began or worsened in severity or relationship to study drug, on or after the date of the first dose of study drug and on or before the date of the last dose of study drug plus 30 days.
  * Had no recorded start date.
Time Frame: 72 weeks
Population: Treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 39 | 41
Percentage of participants | 77 | 85

18. Secondary Outcome: Percentage of Participants Who Discontinue the Study Prematurely (Before Week 48) Due to Adverse Events.
Time Frame: 48 weeks
Population: Treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Zidovudine/Lamivudine
Number analyzed (Participants) | 39 | 41
Percentage of participants | 3 | 10

ADVERSE EVENTS:
Arm/Group | Truvada | Zidovudine/Lamivudine
Serious Adverse Events (participants affected / at risk) | 4 | 3
Other Adverse Events (participants affected / at risk) | 24 | 28
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Truvada | Zidovudine/Lamivudine
Acute myocardial infarction (Cardiac disorders) | 0/39 | 1/41
Prinzmetal angina (Cardiac disorders) | 0/39 | 1/41
Diarrhoea (Gastrointestinal disorders) | 1/39 | 0/41
Respiratory tract infection (Infections and infestations) | 0/39 | 1/41
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1/39 | 0/41
Radius fracture (Injury, poisoning and procedural complications) | 0/39 | 1/41
Cauda equina syndrome (Nervous system disorders) | 1/39 | 0/41
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0/39 | 1/41
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1/39 | 0/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Truvada | Zidovudine/Lamivudine
Anaemia (Blood and lymphatic system disorders) | 1/39 | 3/41
Neutropenia (Blood and lymphatic system disorders) | 0/39 | 3/41
Diarrhoea (Gastrointestinal disorders) | 3/39 | 2/41
Abdominal pain upper (Gastrointestinal disorders) | 2/39 | 0/41
Pyrexia (General disorders) | 2/39 | 0/41
Bronchitis (Infections and infestations) | 2/39 | 0/41
Gamma-glutamyltransferase increased (Investigations) | 11/39 | 10/41
Alanine aminotransferase increased (Investigations) | 8/39 | 10/41
Aspartate aminotransferase increased (Investigations) | 4/39 | 6/41
Blood amylase increased (Investigations) | 4/39 | 8/41
Lipase increased (Investigations) | 1/39 | 3/41
Blood creatine phosphokinase increased (Investigations) | 3/39 | 3/41
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2/39 | 4/41
Hyperlactacidaemia (Metabolism and nutrition disorders) | 2/39 | 0/41
Back pain (Musculoskeletal and connective tissue disorders) | 1/39 | 3/41
Renal colic (Renal and urinary disorders) | 0/39 | 3/41
Blood lactic acid increased (Investigations) | 2/39 | 4/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.